CLINICAL TRIAL: NCT00684398
Title: Adaptation and Quality of Life Among Adults With Neurofibromatosis Type I
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999908144; 08-HG-N144
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2015-11-27

CONDITIONS: Neurofibromatosis Type 1; Von Recklinghausen Disease; NF1
Keywords: Neurofibromatosis Type 1; Quality of Life; Adaptation; Stress and Coping Model; NF1; Survey
MeSH Terms: conditions — Neurofibromatosis 1

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study aims to understand predictors of adaptation and quality of life among adults affected with neurofibromatosis type 1 (NF1) and autosomal dominant neurocutaneous condition. NF1 carries a significant psychosocial burden for affected individuals. Aspects of NF1 that are especially challenging include the unpredictable nature of the disease, variability in severity of symptoms and medical complications, uncertainty in progression, and vulnerability to stigmatization due to the highly visible and often cosmetically disfiguring features of the condition. The literature suggests that because of these and other challenges posed by NF1, affected individuals may struggle to adapt to their condition and, consequently, experience poor quality of life. In this study, Lazarus and Folkman s Tranactional Model of Stress and Coping is used as a framework to conceptualize adaptation and quality of life to NF1. A cross-sectional design with quantitative methodology will be employed to investigate the relationships of appraisals and stigma as predictors of adaptation and quality of life. Adults affected with NF1 will be recruited via regional and national NF organizations and websites, as well as through ongoing NIH clinical research protocols for NF1. Eligible participants will be invited to complete a web-based, self-administered survey....

DETAILED DESCRIPTION:
This study aims to understand predictors of adaptation and quality of life among adults affected with neurofibromatosis type 1 (NF1) and autosomal dominant neurocutaneous condition. NF1 carries a significant psychosocial burden for affected individuals. Aspects of NF1 that are especially challenging include the unpredictable nature of the disease, variability in severity of symptoms and medical complications, uncertainty in progression, and vulnerability to stigmatization due to the highly visible and often cosmetically disfiguring features of the condition. The literature suggests that because of these and other challenges posed by NF1, affected individuals may struggle to adapt to their condition and, consequently, experience poor quality of life. In this study, Lazarus and Folkman s Transactional Model of Stress and Coping is used as a framework to conceptualize adaptation and quality of life to NF1. A cross-sectional design with quantitative methodology will be employed to investigate the relationships of appraisals and stigma as predictors of adaptation and quality of life. Adults affected with NF1 will be recruited via regional and national NF organizations and websites, as well as through ongoing NIH clinical research protocols for NF1. Eligible participants will be invited to complete a web-based, self-administered survey.

ELIGIBILITY:
* INCLUSION CRITERIA:

Adult men and women at least 18 years of age who self-report as having NF1.

Participants must be able to read and write in English.

Individuals of all ethnic, religious, socioeconomic, and educational backgrounds and from a variety of geographic locations in the United States will be included.

EXCLUSION CRITERIA:

Children under the age of 18.

Inability to read and write in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 645 (Actual)
Dates: Start 2008-05-15; Study Completion 2015-11-27

CONTACTS AND LOCATIONS:
Overall Officials: Barbara B Biesecker, Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Radtke HB, Sebold CD, Allison C, Haidle JL, Schneider G. Neurofibromatosis type 1 in genetic counseling practice: recommendations of the National Society of Genetic Counselors. J Genet Couns. 2007 Aug;16(4):387-407. doi: 10.1007/s10897-007-9101-8. Epub 2007 Jul 17. PMID 17636453
- [Background] Ablon J. The nature of stigma and medical conditions. Epilepsy Behav. 2002 Dec;3(6S2):2-9. doi: 10.1016/s1525-5050(02)00543-7. PMID 12609300
- [Background] Benjamin CM, Colley A, Donnai D, Kingston H, Harris R, Kerzin-Storrar L. Neurofibromatosis type 1 (NF1): knowledge, experience, and reproductive decisions of affected patients and families. J Med Genet. 1993 Jul;30(7):567-74. doi: 10.1136/jmg.30.7.567. PMID 8411029